CLINICAL TRIAL: NCT07251309
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 3 Clinical Study to Evaluate the Efficacy and Safety of WS016 in Patients With Hyperkalemia
Brief Title: A Two-Part, Phase 3 Study Evaluating the Efficacy and Safety of WS016 for the Treatment of Hyperkalemia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Waterstone Pharmaceutical (Wuhan) Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WS016CT301
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- WS016 (corrective phase) (Experimental)
  Interventions: Drug: WS016
- Placebo (corrective phase) (Placebo Comparator)
  Interventions: Drug: Placebo
- WS016 (maintenance phase) (Experimental)
  Interventions: Drug: WS016
- Placebo (maintenance phase) (Placebo Comparator)
  Interventions: Drug: Placebo
- WS016 (open-label extension phase) (Experimental)
  Interventions: Drug: WS016

INTERVENTIONS:
Drug: WS016 — WS016 (12g), oral, three times daily for 48 hours, for a total of six doses.
  Arms: WS016 (corrective phase)
Drug: Placebo — Placebo, oral, three times daily for 48 hours, for a total of six doses.
  Arms: Placebo (corrective phase)
Drug: WS016 — WS016 (6g, 12g or 18g), oral, once daily for 28 consecutive days.
  Arms: WS016 (maintenance phase)
Drug: Placebo — Placebo, oral, once daily for 28 consecutive days.
  Arms: Placebo (maintenance phase)
Drug: WS016 — WS016, oral, once daily for 11 months, starting at a dose of 12g with subsequent dose adjustments based on serum potassium levels.
  Arms: WS016 (open-label extension phase)

SUMMARY:
This clinical trial consists of 2 parts, Part A and Part B. Part A consists of a 2-day randomized, double-blind, placebo-controlled corrective phase (CP) and a 28-day randomized, double-blind, placebo-controlled maintenance phase (MP). Part B (open-label extension, OLE) is an open-label, 11-month extension study carried out in participants who come from Part A and meet certain inclusion criteria.

DETAILED DESCRIPTION:
Eligible participants with hyperkalemia will first be randomized in a 5:1 ratio to receive oral WS016 (12g) or placebo three times daily, for a total of six doses over 48 hours.

After the 48-hour corrective treatment, participants whose serum potassium is within the normal range will be re-randomized in a 1:1:1:1 ratio to receive oral WS016 (6g, 12g, or 18g) or placebo once daily for 28 consecutive days.

Participants who complete the 28-day maintenance phase or prematurely discontinue from it due to hyperkalemia or hypokalemia, and who meet the eligibility criteria, will be eligible to enter Part B. In Part B, participants will receive WS016 for 11 months, starting at 12g once daily, with subsequent dose adjustments based on serum potassium levels.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male or female) aged 18 years and older;
* Participants with a serum potassium concentration >5.0 mmol/L and ≤6.5 mmol/L (serum potassium concentration will be measured using the i-STAT portable biochemical analyzer in screening period);
* Participants who have negative pregnancy test result at screening and ensure the use of contraception during the trial;
* Participants who understand and voluntarily sign the Informed Consent Form.

Exclusion Criteria:

* Participants who have a history of severe drug allergy, or are definitely allergic to the investigational product or its ingredients;
* Participants who have pseudohyperkalemia, such as serum potassium increasing caused by hemolysis of blood samples due to improper blood collection methods (such as too tight pressure pulse band banding, too heavy local rubbing, repeated fist clenching-loosening hands), hemolysis of blood samples due to difficulty in venipuncture or trauma, and severe leukocytosis (>50 × 10^9/L) or thrombocytosis (>500 × 10^9/L);
* Participants with acute hyperkalemia caused by conditions such as tumor lysis syndrome or hemolysis and so on;
* Participants suffering from severe cerebrovascular diseases, such as cerebral infarction or cerebral hemorrhagic disease, with language disorder or unresponsiveness, or severely blocked limb movement;
* Participants who have suffered from myocardial infarction, or have undergone interventional cardiac procedures or coronary artery bypass grafting for coronary atherosclerotic heart disease within 3 months prior to screening; or participants who have heart failure and are in cardiac function class IV (New York Heart Association, NYHA classification criteria) at screening;
* Participants with cardiac arrhythmia requiring urgent treatment at screening, such as ventricular tachycardia, ventricular fibrillation, II-III degree atrioventricular block, severe bradycardia (heart rate <40 bpm), or participants with significant prolongation of PR interval (PR interval prolonged to more than 0.25 seconds in the absence of pre-existing atrioventricular block), decrease or disappearance of P wave amplitude, and widening of QRS wave (widening to more than 0.14 seconds in the absence of pre-existing bundle branch block) indicated by the electrocardiogram at screening;
* Participants who have previously undergone major gastrointestinal surgery such as subtotal gastrectomy, short bowel syndrome and other diseases affecting the normal peristalsis of the gastrointestinal tract; or participants with intractable constipation;
* Participants who have received treatment with polypropylene exchange resin or sodium zirconium cyclosilicate and other similar drugs within 3 days before screening;
* Participants who participated in other clinical trials of drugs or devices not approved for marketing within 3 months prior to the first dose;
* Participants who are receiving dialysis;
* Participants with severe hepatic impairment: serum alanine aminotransferase or aspartate aminotransferase more than 3 times the upper limit of normal;
* Participants who are unable to complete this part of the trial as assessed by the investigator due to any other disease or psychiatric condition; or participants whose participation in the trial is assessed by the investigator as having a risk that far outweighs the benefit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Mean serum potassium level during maintenance phase Days 8-29 | Maintenance phase Days 8-29

SECONDARY OUTCOMES:
Exponential rate of change in serum potassium during the corrective phase | Through 48 hours corrective phase
Mean change from baseline in serum potassium at all time points of corrective phase | Through 48 hours corrective phase
Cumulative duration (in days) of serum potassium within the normal range during the maintenance phase | Maintenance phase baseline to maintenance phase Day 29
Mean change from baseline in serum potassium at all time points of maintenance phase | Through 28 days maintenance phase
Percentage of participants with the mean serum potassium ≤5.0 mmol/L and percentage of participants with the mean serum potassium ≤5.5 mmol/L from D8 to D337 of the open-label extension phase | Open-label extension phase Days 8-337

CONTACTS AND LOCATIONS:
Locations (50):
- China (50):
  - Investigator Site 02, Bengbu, Anhui
  - Investigator Site 03, Wuhu, Anhui
  - Investigator Site 48, Chongqing, Chongqing Municipality
  - Investigator Site 04, Xiamen, Fujian
  - Investigator Site 05, Lanzhou, Gansu
  - Investigator Site 07, Guangzhou, Guangdong
  - Investigator Site 06, Zhanjiang, Guangdong
  - Investigator Site 08, Huizhou, Guangxi
  - Investigator Site 09, Nanning, Guangxi
  - Investigator Site 10, Nanning, Guangxi
  - Investigator Site 11, Guiyang, Guizhou
  - Investigator Site 12, Haikou, Hainan
  - Investigator Site 13, Shijiazhuang, Hebei
  - Investigator Site 18, Daqing, Heilongjiang
  - Investigator Site 15, Nanyang, Henan
  - Investigator Site 16, Nanyang, Henan
  - Investigator Site 14, Puyang, Henan
  - Investigator Site 25, Xinxiang, Henan
  - Investigator Site 21, Huangshi, Hubei
  - Investigator Site 20, Shiyan, Hubei
  - Investigator Site 19, Wuhan, Hubei
  - Investigator Site 22, Wuhan, Hubei
  - Investigator Site 24, Hengyang, Hunan
  - Investigator Site 17, Yueyang, Hunan
  - Investigator Site 23, Zhuzhou, Hunan
  - Investigator Site 37, Chifeng, Inner Mongolia
  - Investigator Site 36, Hohhot, Inner Mongolia
  - Investigator Site 30, Changzhou, Jiangsu
  - Investigator Site 31, Huai'an, Jiangsu
  - Investigator Site 01, Nanjing, Jiangsu
  - Investigator Site 26, Nantong, Jiangsu
  - Investigator Site 27, Suzhou, Jiangsu
  - Investigator Site 29, Yangzhou, Jiangsu
  - Investigator Site 32, Ganzhou, Jiangxi
  - Investigator Site 33, Nanchang, Jiangxi
  - Investigator Site 34, Shangrao, Jiangxi
  - Investigator Site 35, Shenyang, Liaoning
  - Investigator Site 38, Yinchuan, Ningxia
  - Investigator Site 42, Xi'an, Shaanxi
  - Investigator Site 43, Xi'an, Shaanxi
  - Investigator Site 41, Jinan, Shandong
  - Investigator Site 40, Qingdao, Shandong
  - Investigator Site 39, Tancheng, Shandong
  - Investigator Site 44, Shanghai, Shanghai Municipality
  - Investigator Site 45, Chengdu, Sichuan
  - Investigator Site 47, Chengdu, Sichuan
  - Investigator Site 46, Deyang, Sichuan
  - Investigator Site 49, Zigong, Sichuan
  - Investigator Site 28, Jiaxing, Zhejiang
  - Investigator Site 50, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No